CLINICAL TRIAL: NCT03085472
Title: Chongqing Intracerebral Hemorrhage Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qi Li, Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: X1517
Record Dates: First submitted 2017-03-01; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Intracerebral Hemorrhage; Stroke; Hematoma
Keywords: intracerebral hemrrohage; stroke; China; hematoma; CT; predictor; prognosis; outcome
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hematoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- benigh hematoma: Patients with novel imaging markers or clinical features suggestive of a relatively benigh hematoma (less likely to expand and have a relatively good outcome).
- malignant hematoma: Patients with novel imaging markers or clinical features suggestive of a relatively bad hematoma (more likely to expand and have a relatively poor outcome).

SUMMARY:
The Chongqing intracerebral hemorrhage study is a multi-center, prospective, observational study led by professor Qi Li from Chongqing Medical University. Professor Peng Xie will be the senior consultant for the study. The Chongqing intracerebral hemorrhage study will focus on the epidemiology, natural history, pathogenesis, laboratory, radiological aspects, clinical outcomes and the effects of treatment in patients with intracerebral hemorrhage.

The clinical, laboratory, imaging, genetic and outcome data of patients diagnosed with acute intracerebral hemorrhage will be prospectively collected. The prognosis of patients with intracerebral hemorrhage will be assessed by using several outcome measure scales at different time points.

DETAILED DESCRIPTION:
The Chongqing intracerebral hemorrhage study will try to address several key issues in ICH. The baseline clinical data including demographic, disease severity scores, prior drug history and relevant medical history, premorbid mRS scores will be prospectively recorded. The admission and follow-up imaging data of all registered patients will be saved as Dicom format for future use and review. The functional outcomes will be assessed and recorded by experienced neurologists.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Informed consent to participate in the study
* Patients diagnosed with CT-confirmed spontaneous Intracerebral Hemorrhage (ICH)
* Patients are willing to participate in the follow up assessment

Exclusion Criteria:

* Did not agree to participate in the study
* Secondary ICH to hemorrhagic infarction or tumor bleeding etc.
* Traumatic ICH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 Years and older (Adult patients)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
hematoma volume growth at 24 hours | 24 hours
  To assess early hematoma volume growth at 24 hours

SECONDARY OUTCOMES:
functional outcome at 3 months assessed by modified Ranking Scale | 3 months
  assess functional outcome at 3months using mRS
early neurological deterioration assessed by NIHSS score at 24 hours | 24 hours
  To assess early neurological deterioration using NIHSS score at 24 hours
early neurological deterioration assessed by NIHSS at 48 hours | 48 hours
  To assess early neurological deterioration using NIHSS score at 48 hours
early neurological deterioration assessed by NIHSS score | 72hours
  To assess early neurological deterioration using NIHSS score at 72 hours
perihematoma edema volume measurement at 24 hours | 24 hours
  to measure the perihematoma edema volume at 24 hours
perihematoma edema volume measurement at 72 hours | 72 hours
  to measure the perihematoma edema volume at 72 hours
intraventricular hemorrhage growth | 24 hours
  to assess the presence of IVH at 24 hours
major thromboembolic events | 2 weeks
  to assess the thromboembolic events 2 weeks after admission

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided